CLINICAL TRIAL: NCT01450579
Title: Phase II Study of ASP7373 Evaluation of Immunogenicity and Safety of ASP7373 in Healthy Adults
Brief Title: A Study to Evaluate the Immune Response to the ASP7373 and Its Safety in Healthy Adult Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMN Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 7373-CL-0106
Record Dates: First submitted 2011-09-22; First posted 2011-10-12 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Recombinant Influenza HA vaccine; Immunogenicity of ASP7373

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Saline
  Interventions: Biological: Placebo
- Dose -1 (Experimental): ASP7373
  Interventions: Biological: ASP7373
- Dose -2 (Experimental): ASP7373
  Interventions: Biological: ASP7373
- Dose -3 (Experimental): ASP7373
  Interventions: Biological: ASP7373

INTERVENTIONS:
Biological: ASP7373 — Intermuscular administration
  Arms: Dose -1; Dose -2; Dose -3
Biological: Placebo — Intramuscular administration
  Arms: Placebo

SUMMARY:
This trial is to investigate the clinically recommended dosage for ASP7373 based on the comparison of the immunogenicity and safety among the three doses of ASP7373 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: Female: ≥40.0 kg, <70.0 kg, Male: ≥50.0 kg, <80.0 kg
* BMI: ≥17.6, <26.4
* Healthy, as judged by the investigator or sub-investigator based on the results of physical examinations (subjective symptoms and objective findings) and all tests obtained

Exclusion Criteria:

* Scheduled to receive another vaccine during study period
* History of H5 influenza infection or received H5 influenza vaccine
* Past history of anaphylactic shock or an allergic reaction such as generalized eruption due to food or drug (including vaccines) allergies, fever ≥ 39.0°C within 2 days after the previous vaccination (influenza vaccine and others)
* Diagnosis of immune deficit in the past, has a family member (within the third degree of kinship) with a diagnosis of congenital immunodeficiency syndrome
* Received or scheduled to receive a live vaccine within 28 days prior to vaccination of the study vaccine, and received or scheduled to receive an inactivated vaccine or a toxoid within 7 days prior to vaccination of the study vaccine
* History of seizures
* Female subjects who are breastfeeding, pregnant, possibly pregnant, and planning to become pregnant during the study period

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety assessed by the incidence of adverse events, vital signs, laboratory tests and 12-lead ECGs | up to 43 days
Immunogenicity (HI antibody titer)- first vaccine | on Day 21
Immunogenicity (HI antibody titer)- second vaccine | on Day 43
  second vaccination on Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan